CLINICAL TRIAL: NCT02802657
Title: A Multicenter Study Comparing Efficacy and Safety of " Treat-and-Extend" Regimen Versus "Pro Re Nata" Regimen of Conbercept in Neovascular Age-related Macular Degeneration
Brief Title: Efficacy and Safety of "Treat-and-Extend" Regimen Versus "Pro Re Nata" of Conbercept in Age-related Macular Degeneration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiaodong Sun (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other); Shanghai Zhongshan Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); The General Hospital of Central Theater Command (Other)
Responsible Party: Sponsor-Investigator, Xiaodong Sun, Professor and Executive Vicechair of Department of Ophthalmology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15216713049
Record Dates: First submitted 2016-06-05; First posted 2016-06-16 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related Macular Degeneration; Conbercept; Treat-and-Extend Regimen; Pro Re Nata
MeSH Terms: conditions — Macular Degeneration | interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conbercept 0.5mg Treat-and-Extend regimen (Experimental): Monthly intravitreal injections of Conbercept 0.5mg in the core treatment period and Treat-and-Extend Regimen of the same dose guided by BCVA stabilization and optical coherence tomography (OCT) in the extension treatment period.
  Intervention: Drug: Conbercept
  Interventions: Procedure: Treat-and-Extend regimen; Drug: Conbercept
- Conbercept 0.5mg Pro Re Nata (Active Comparator): Monthly intravitreal injections of Conbercept 0.5mg in the core treatment period and PRN intravitreal injections of the same dose guided by BCVA stabilization in the extension treatment period.
  Intervention: Drug: Conbercept
  Interventions: Procedure: Pro Re Nata; Drug: Conbercept

INTERVENTIONS:
Procedure: Treat-and-Extend regimen — For the T&E regimen,investigators recorded patients' data after retreatment by 3 monthly intravitreal injections of Conbercept. Patients were examined 6 weeks after the third injection, with ETDRS visual acuity testing, fundus ophthalmoscopy and photography, and OCT, and treated on the same day. The interval between treatments was extended by 2-week (12-week was a maximum) provided that OCT and fundus examination did not show either exudative manifestations or new macular hemorrhage or active CNV or reduced by 2 weeks (4-week was minimum) in case of such manifestations or hemorrhage. The persistence of pigment epithelium detachment was not considered a condition that justified shortening the interval between injections.
  Other Names: T&E
  Arms: Conbercept 0.5mg Treat-and-Extend regimen
Procedure: Pro Re Nata — For the PRN group, investigators recorded patients'data after retreatment by 3 monthly intravitreal injections of Conbercept.Subsequent reinjections were given as needed according to the changes in patients'visual acuity and/or the exudation shown by OCT. Four to five weeks after the third and last injection, all patients in the PRN group underwent an examination, including ETDRS visual acuity, fundus photography,and OCT. In case of persistent subfoveal or perifoveal fluid, macular intraretinal edema, visual loss of >5 letters, or the occurrence of a new hemorrhage, patients were retreated. The persistence of hemorrhage without evidence of fluid was not considered a criterion for retreatment. In the absence of retreatment criteria, no further injections were given and another examination was proposed usually 4 weeks later.
  Other Names: PRN
  Arms: Conbercept 0.5mg Pro Re Nata
Drug: Conbercept

SUMMARY:
The study will evaluate the efficacy and safety of two different regimens of Conbercept (Treat-and-Extend (T&E) Regimen vs. Pro Re Nata (PRN)) in patients with wet AMD. This study is to provide long-term safety data in the treatment of patients with wet Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
Participants with wAMD were randomized and received a T&E or PRN regimen for 24 months. Mean Snellen BCVA and mean central macular thickness by OCT were examined at each visit. Any treatment-related adverse events, such as endophthalmitis, and systemic adverse events, such as stroke, were evaluated during the research.

ELIGIBILITY:
Inclusion Criteria:

* Written informed-consent before any evaluation
* Visual impairment due to active CNV,including predominantly classic CNV,minimally classic CNV,occult CNV with no classic component and PCV.
* 50 years old and older
* Chinese
* For study eye: BCVA between 20/30 and 20/320 on electronic visual acuity texting at the time point of both screening and baseline.

Exclusion Criteria:

* Have Stroke and myocardial infarction within 3 months before screening
* Any active periocular and ocular infection and inflammation (including blepharitis, conjunctivitis, keratitis, scleritis, uveitis, intraocular inflammation) while screening and baseline.
* Uncontrolled glaucoma (under treatment [IOP] ≥ 30 mm Hg or depend on researchers) while screening and baseline
* Neovascularization of iris and neovascular glaucoma while screening and baseline
* Any causes led to choroidal neovascularization except Wet AMD (including ICNV,central serous chorioretinopathy,ocular histoplazmoza and pathologic myopia) while screening and baseline
* With structure injury (including vitreous macular traction,epiretinal membrane involving in central fovea,subretinal fibroplasia,laser scar and central fovea atrophy) within 0.5 optic disc diameter to the central of macula while screening and baseline, which may harm the improvement of vision by treatment according to researchers
* Any systemic anti-VEGF medication(as Avastin) use within 3 months before screening
* Any medication systemic use toxic to lens, retina and optic nerve,including iron amine, chloroquine/chloroquine (Plaquenil ®), tamoxifen, phenothiazine and ethambutol
* For study eye：Used to accept following treatments for wet AMD within 3 months or accept following treatments more than three times before baseline: a)Anti-angiogenesis drugs(pegaptanib （Macugen®），ranibizumab ,bevacizumab（Avastin®),VEGF-Trap，KH902；b）Anecortave acetate corticosteroids；c）Protein kinase C inhibitors，squalamine，siRNA; d)PDT （Visudyne®）treatment,external beam radiotherapy, local laser photocoagulation, vitrectomy, submacular surgery and transpupillary thermotherapy
* Any intraocular surgery(including YAG laser) within 3 months before baseline or predicated within 6 months after baseline
* Intraocular or periocular treatment of corticosteroids within 3 months before baseline
* For follow eye:Any anti-angiogenesis treatment(including anti-VEGF,like Lucentis,Avastin® and KH902 ) within 3 months before baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Mean Snellen BCVA at every visit or treatment | 24 months
  Compare of mean Snellen Best-Corrected-visual-acuity at every visit or treatment between the two groups to assess the efficacy of Treat-and-Extend regimen of Conbercept.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 24 months
  Compare of Number of participants with treatment-related adverse events between the two groups to assess the safety of Treat-and-Extend regimen of Conbercept
Mean number of injections after the initial three loading dose monthly injections | 21 months
  Compare of mean number of injections after the initial three loading dose monthly injections between the two groups to assess the efficacy of Treat-and-Extend regimen of Conbercept.
mean central macular thickness at every visit or treatment by OCT | 24 months
  Compare of mean central macular thickness by OCT at every visit or treatment between the two groups to assess the efficacy of Treat-and-Extend regimen of Conbercept.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University
Locations (5):
- China (5):
  - Central Theater Command General Hospital, Wuhan, Hubei
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rush RB, Simunovic MP, Vandiver L, Aragon AV 2nd, Ysasaga JE. Treat-and-extend bevacizumab for neovascular age-related macular degeneration: the importance of baseline characteristics. Retina. 2014 May;34(5):846-52. doi: 10.1097/IAE.0000000000000033. PMID 24240560
- [Background] Chen YN, Powell AM, Mao A, Sheidow TG. RETROSPECTIVE REVIEW OF LUCENTIS "TREAT AND EXTEND" PATTERNS AND OUTCOMES IN AGE-RELATED MACULAR DEGENERATION. Retina. 2016 Feb;36(2):272-8. doi: 10.1097/IAE.0000000000000691. PMID 26200511
- [Background] Wykoff CC, Croft DE, Brown DM, Wang R, Payne JF, Clark L, Abdelfattah NS, Sadda SR; TREX-AMD Study Group. Prospective Trial of Treat-and-Extend versus Monthly Dosing for Neovascular Age-Related Macular Degeneration: TREX-AMD 1-Year Results. Ophthalmology. 2015 Dec;122(12):2514-22. doi: 10.1016/j.ophtha.2015.08.009. Epub 2015 Sep 29. PMID 26391465
- [Background] Spaide R. Ranibizumab according to need: a treatment for age-related macular degeneration. Am J Ophthalmol. 2007 Apr;143(4):679-80. doi: 10.1016/j.ajo.2007.02.024. No abstract available. PMID 17386275
- [Background] Mrejen S, Jung JJ, Chen C, Patel SN, Gallego-Pinazo R, Yannuzzi N, Xu L, Marsiglia M, Boddu S, Freund KB. Long-Term Visual Outcomes for a Treat and Extend Anti-Vascular Endothelial Growth Factor Regimen in Eyes with Neovascular Age-Related Macular Degeneration. J Clin Med. 2015 Jul 8;4(7):1380-402. doi: 10.3390/jcm4071380. PMID 26239682
- [Background] Berg K, Hadzalic E, Gjertsen I, Forsaa V, Berger LH, Kinge B, Henschien H, Fossen K, Markovic S, Pedersen TR, Sandvik L, Bragadottir R. Ranibizumab or Bevacizumab for Neovascular Age-Related Macular Degeneration According to the Lucentis Compared to Avastin Study Treat-and-Extend Protocol: Two-Year Results. Ophthalmology. 2016 Jan;123(1):51-9. doi: 10.1016/j.ophtha.2015.09.018. Epub 2015 Oct 21. PMID 26477842
- [Background] Oubraham H, Cohen SY, Samimi S, Marotte D, Bouzaher I, Bonicel P, Fajnkuchen F, Tadayoni R. Inject and extend dosing versus dosing as needed: a comparative retrospective study of ranibizumab in exudative age-related macular degeneration. Retina. 2011 Jan;31(1):26-30. doi: 10.1097/IAE.0b013e3181de5609. PMID 20890246
- [Background] Chin-Yee D, Eck T, Fowler S, Hardi A, Apte RS. A systematic review of as needed versus treat and extend ranibizumab or bevacizumab treatment regimens for neovascular age-related macular degeneration. Br J Ophthalmol. 2016 Jul;100(7):914-917. doi: 10.1136/bjophthalmol-2015-306987. Epub 2015 Oct 29. PMID 26516125
- [Background] Houston SK 3rd, Rayess N, Cohen MN, Ho AC, Regillo CD. INFLUENCE OF VITREOMACULAR INTERFACE ON ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR THERAPY USING TREAT AND EXTEND TREATMENT PROTOCOL FOR AGE-RELATED MACULAR DEGENERATION (VINTREX). Retina. 2015 Sep;35(9):1757-64. doi: 10.1097/IAE.0000000000000663. PMID 26110596
- [Background] Gupta OP, Shienbaum G, Patel AH, Fecarotta C, Kaiser RS, Regillo CD. A treat and extend regimen using ranibizumab for neovascular age-related macular degeneration clinical and economic impact. Ophthalmology. 2010 Nov;117(11):2134-40. doi: 10.1016/j.ophtha.2010.02.032. Epub 2010 Jul 1. PMID 20591490
- [Background] Abedi F, Wickremasinghe S, Islam AF, Inglis KM, Guymer RH. Anti-VEGF treatment in neovascular age-related macular degeneration: a treat-and-extend protocol over 2 years. Retina. 2014 Aug;34(8):1531-8. doi: 10.1097/IAE.0000000000000134. PMID 24637667
- [Background] Homer N, Grewal DS, Mirza RG, Lyon AT, Gill MK. Transitioning to intravitreal aflibercept following a previous treat-and-extend dosing regimen in neovascular age-related macular degeneration: 24-month results. Eye (Lond). 2015 Sep;29(9):1152-5. doi: 10.1038/eye.2015.87. Epub 2015 May 29. PMID 26021870
- [Background] Li X, Xu G, Wang Y, Xu X, Liu X, Tang S, Zhang F, Zhang J, Tang L, Wu Q, Luo D, Ke X; AURORA Study Group. Safety and efficacy of conbercept in neovascular age-related macular degeneration: results from a 12-month randomized phase 2 study: AURORA study. Ophthalmology. 2014 Sep;121(9):1740-7. doi: 10.1016/j.ophtha.2014.03.026. Epub 2014 May 1. PMID 24793528
- [Background] Zhang M, Zhang J, Yan M, Luo D, Zhu W, Kaiser PK, Yu DC; KH902 Phase 1 Study Group. A phase 1 study of KH902, a vascular endothelial growth factor receptor decoy, for exudative age-related macular degeneration. Ophthalmology. 2011 Apr;118(4):672-8. doi: 10.1016/j.ophtha.2010.08.008. Epub 2010 Dec 13. PMID 21146224
- [Derived] Jia H, Lu B, Yuan Y, Yuan F, Li L, Song Y, Rong A, Zhou M, Wang F, Sun X. A Randomized, Controlled Trial of Treat-and-Extend vs. Pro Re Nata Regimen for Neovascular Age-Related Macular Degeneration. Front Med (Lausanne). 2022 Jun 20;9:852519. doi: 10.3389/fmed.2022.852519. eCollection 2022. PMID 35795633